CLINICAL TRIAL: NCT03993301
Title: The Impact of Infant Formula With Probiotics on Infants Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Glac Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Hung-Chih Lin, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMUH108-REC2-005
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-03

CONDITIONS: Probiotics Infant Formula; Infants Health
Keywords: Probiotics; Infant formula; Gastroenteritis; Allergy; Respiratory infection
MeSH Terms: conditions — Gastroenteritis; Hypersensitivity; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic A formula (Experimental): Infant Formula with Lactobacillus salivarius AP-32
  Interventions: Other: Probiotic A formula
- Probiotic B formula (Experimental): Infant Formula with Bifidobacterium animalis subsp. lactis CP-9
  Interventions: Other: Probiotic B formula
- Regular formula (Placebo Comparator): The infant formula without any probiotic.
  Interventions: Other: Regular formula

INTERVENTIONS:
Other: Probiotic A formula — Feeding baby two meals a day with Infant formula with probiotics (10^8 colony-forming unit per day) at least.
  Arms: Probiotic A formula
Other: Probiotic B formula — Feeding baby two meals a day with Infant formula with probiotics (10^8 colony-forming unit per day) at least.
  Arms: Probiotic B formula
Other: Regular formula — Feeding baby two meals a day with regular formula at least.
  Arms: Regular formula

SUMMARY:
The trial will be divided into three groups, the experimental group: (I) probiotic A formula, (II) probiotic B formula; control group: (III) regular formula (Youluck infant formula). Inclusion criteria included: (1) the normal spontaneous delivery (NSD) full-term health infants (≧37 weeks) and birth weight more than 2500 grams and (2) subjects who are expected to breastfeed are eligible for the trial after informed consent form is signed by the parents. Exclusion criteria included: infants with chronic diarrhea, hemangioma, cerebral hemorrhage, severe asphyxia (stage III), fetal chromosomal abnormalities, cyanotic congenital heart disease, intestinal hypoplasia or abnormal immune function after birth, liver failure, breastfeeding within two months after birth, taking other probiotic products within two weeks after birth, treatment with antibiotics during acute infection and diagnosis of allergies, gastroenteritis, respiratory infections will be excluded. The study will be conducted for half a year, 5 cans of Youluck infant formula are provided for each subject during the test period. The Youluck infant formula is sponsored free of charge by glac biotech Co., Ltd. During hospitalization, the infant will be feed by same group of experienced nurses and all infants will be monitored for adverse conditions such as vomiting, diarrhea or bloating every day.

DETAILED DESCRIPTION:
Probiotics were defined as an ''live microorganisms, which, when administered in adequate amounts, conferred a health benefit on the host. Before 2005, some animal experiments indicated that probiotics could help weight gain. In 2006, there was a team observed the growth of infants who received infant formula with probiotics. The study found that infants who received infant formula with probiotics for half a year had higher height and weight than infants who received regular formula, and the defecation frequency was increased. So far, clinical studies had proved that probiotics had an efficacy on gastrointestinal immune regulation. Some studies had found that concentrated preparations mixed with various probiotics had therapeutic effects on inflammatory bowel diseases. The latest double-blind study of infants with acute diarrhoea showed that oral dehydration supplements enriched probiotics and zinc could reduce the severity of diarrhoea on day 2 without any side effects. Therefore, more and more probiotic clinical studies had suggested that probiotics could be used to regulate gastrointestinal related diseases.

According to statistics, the proportion of atopic dermatitis in infants and children worldwide is about 10-20%, and about 30% of toddlers with more than three episodes of wheezing bronchitis may develop persistent asthma. Therefore, how to effectively prevent the occurrence of allergic diseases was still an urgent goal for infants and young children. There is now evidence in mice and humans of an early-life "critical window" in which the effects of gut microbial dysbiosis are most influential in human immune development. Investigators showed that infants at risk of asthma exhibited transient gut microbial dysbiosis during the first 100 days of life. Inoculation of the relatively lower abundance of the genus to asthmatic mice ameliorated airway inflammation. These results enhanced the potential for future microbe-based diagnostics and therapies, potentially in the form of probiotics, to prevent the development of asthma and other related allergic diseases in children.

In addition, respiratory infections were diseases that needed attention during the growth phase of infants and young children. The most common treatment for respiratory infections or acute otitis media in infants and young children was using antibiotics, but antibiotic treatment might lead to antibiotic resistance and intestinal microbial disorders, which might promote colonization of pathogens. In recent years, probiotics had attracted more and more attention for the prevention of respiratory infections. For example, investigators showed that using Bifidobacterium probiotics in children before 2 years old might reduce the incidence of respiratory infections.

Based on the above studies, Investigators will use infant formula with probiotics to infants. The study will assess the growth, incidence of allergies, gastroenteritis and respiratory infections of infants. This observational study will be conducted at the China Medical University Children's Hospital performed a double-blind randomized trial.

The trial will be divided into three groups, the experimental group: (I) probiotic A formula, (II) probiotic B formula; control group: (III) regular formula (Youluck infant formula). Inclusion criteria included: (1) the normal spontaneous delivery (NSD) full-term health infants (≧37 weeks) and birth weight more than 2500 grams and (2) subjects who are expected to breastfeed are eligible for the trial after informed consent form is signed by the parents. Exclusion criteria included: infants with chronic diarrhea, hemangioma, cerebral hemorrhage, severe asphyxia (stage III), fetal chromosomal abnormalities, cyanotic congenital heart disease, intestinal hypoplasia or abnormal immune function after birth, liver failure, breastfeeding within two months after birth, taking other probiotic products within two weeks after birth, treatment with antibiotics during acute infection and diagnosis of allergies, gastroenteritis, respiratory infections will be excluded. The study will be conducted for half a year, 5 cans of Youluck infant formula are provided for each subject during the test period. The Youluck infant formula is sponsored free of charge by glac biotech Co., Ltd. During hospitalization, the infant will be feed by same group of experienced nurses and all infants will be monitored for adverse conditions such as vomiting, diarrhea or bloating every day. After the study is completed, the remaining probiotic milk powder will be subjected to high temperature and high pressure for sterilization, and then placed in an infectious garbage bag or infective trash can, and destructed by a cleaning company.

Sample size calculation is based on the literature. The incidence of enteritis, allergic disease or respiratory infection in infants is about 30%. Investigators assume that the experimental group has a 50% improvement compared with the control group. If investigators allow 5% chance of type 1 error (α=0.05) and 10% chance of type 2 error (β=0.1), then the required sample size in each group will be 60 people (total 180 infants in three groups).

The research data will be based on International Business Machines Statistical Product and Service Solutions (IBM SPSS) for analytical statistics. Normally distributed data were analyzed using Student's t-test two-tailed assay, and non-normally distributed data were analyzed using the Wilcoxon signed-rank test. Data were presented as mean ± standard deviation (SEM) or median, with P values < 0.05 being considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. The normal spontaneous delivery (NSD) full-term health infants (≧37 weeks) and birth weight more than 2500 grams.
2. Subjects who are expected to breastfeed are eligible for the trial after informed consent form is signed by the parents.

Exclusion Criteria:

1. Chronic diarrhea
2. Hemangioma
3. Cerebral hemorrhage
4. Severe asphyxia (stage III)
5. Fetal chromosomal abnormalities
6. Cyanotic congenital heart disease
7. Intestinal hypoplasia or abnormal immune function after birth.
8. Liver failure
9. Breastfeeding within two months after birth.
10. Taking other probiotic products within two weeks after birth.
11. Treatment with antibiotics during acute infection and diagnosis of allergies.
12. Gastroenteritis
13. Respiratory infections

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 6 month follow-up.
  All babies are monitored for adverse events such as vomiting, diarrhea or bloating.
Change in body weight | 6 month follow-up.
  The baby will record the body weight before taking infant formula. During the half-year trial period, the body weight will also be measured every 2 months.
Change in body height | 6 month follow-up.
  The baby will record the body height before taking infant formula. During the half-year trial period, the body height will also be measured every 2 months.
Change in head circumference | 6 month follow-up.
  The baby will record the head circumference before taking infant formula. During the half-year trial period, the head circumference will also be measured every 2 months.

SECONDARY OUTCOMES:
The occurrence of inflammatory bowel diseases | 6 month follow-up.
The occurrence of allergic diseases | 6 month follow-up.
The occurrence of respiratory infection | 6 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chih Lin, Principal Investigator — China Medical University Hospital
Locations (1):
- Department of Pediatrics, Children Hospital, China Medical University, Taichung, Taiwan

REFERENCES:
- [Derived] Shen SP, Lin HC, Chen JF, Wang HS, Huang YY, Hsia KC, Lin JH, Kuo YW, Li CM, Hsu YC, Tsai SY, Ho HH. Assessment of the safety and gut microbiota modulation ability of an infant formula containing Bifidobacterium animalis ssp. lactis CP-9 or Lactobacillus salivarius AP-32 and the effects of the formula on infant growth outcomes: insights from a four-month clinical study in infants under two months old. BMC Pediatr. 2024 Dec 27;24(1):840. doi: 10.1186/s12887-024-05289-7. PMID 39731060